CLINICAL TRIAL: NCT03324126
Title: Effects of Targeted Versus Adjustable Protein Fortification of Breast Milk on Early Growth in Very-low-birth-weight Preterm Infants: A Randomized Clinical Trial
Brief Title: Individualized Fortification of Breast Milk
Status: Completed | Type: Observational
Sponsor: Ozgul Bulut (Other)
Responsible Party: Sponsor-Investigator, Ozgul Bulut, Principal Investigator, Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: 35496
Record Dates: First submitted 2017-09-30; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Breast Milk; Premature Infant
Keywords: Preterm infants; very low birth weight; breast milk; individualized fortification; targeted protein fortification; adjustable protein fortification; growth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Targeted fortification: In the targeted protein fortification group, breast milk samples were analyzed daily via mid-infrared spectroscopy and additional protein was provided to maintain an intake of 4.5 g/kg/day.
- Adjustable fortification: In the adjustable protein fortification group, blood urea nitrogen (BUN) levels were monitored weekly, and if the level was < 5 mg/dL, the amount of protein fortification was gradually increased to an "estimated" maximum level of 4.5 g/kg/day

SUMMARY:
Objectives: To compare the effects of two different methods of individualized protein fortification of breast milk on the early growth of VLBW preterm infants.

Design: VLBW preterm infants ≤ 32 weeks of gestational age were included in the study and randomized into two groups according to the method of breast milk fortification. In the targeted protein fortification group, breast milk samples were analyzed daily via mid-infrared spectroscopy and additional protein was provided to maintain an intake of 4.5 g/kg/day. In the adjustable protein fortification group, blood urea nitrogen (BUN) levels were monitored weekly, and if the level was < 5 mg/dL, the amount of protein fortification was gradually increased to an "estimated" maximum level of 4.5 g/kg/day, as per the policy of neonatal intensive care unit. The cumulative amounts of protein, energy, fat, and carbohydrate given to infants prior to study commencement and during the study period were calculated. Anthropometric measurements were performed in both groups weekly for 4 weeks to compare their growth, and blood data including pH, base deficit, and urea, creatinine, and albumin levels were collected.

DETAILED DESCRIPTION:
Optimal feeding during the early neonatal period is critical because inadequate nutrition, especially of very-low-birth-weight (VLBW) preterm infants, causes growth restrictions and has negative effects on neurocognitive development (1-5).

Although breast milk is the first choice for nutrition of preterm infants (6, 7), it falls short of meeting all of the nutritional needs of VLBW infants unless fortified (8-10). Therefore, standard fortification (addition of a fixed amount of a commercial fortifier to breast milk) has become a commonly used method in neonatal intensive care units (NICUs) (11, 12). Standard fortification is performed based on assumptions made about the protein level in breast milk. However, protein levels show inter- and intra-individual variation, and the assumed levels in the milk of the mothers of preterm infants (2.1-2.4 g/100 kcal) is reduced to <1.5 g/100 kcal after the 14th day of lactation (10, 13-17). The protein content of commercial fortifiers ranges from 0.7 to 1.1 g/100 mL, and they thus can only increase the amount of protein in breast milk to 3.25 g/100 kcal. Therefore, the standard fortification method fails to meet the daily protein need of 3.5-4.5 g/kg/day of VLBW infants that is recommended by the European Society for Pediatric Gastroenterology Hepatology and Nutrition (18, 19).

Individualized fortification is another method recommended for optimizing breast milk fortification, and it is considered the best solution for addressing the protein deficiencies of VLBW preterm infants (10, 12). There are two valid methods of individualized fortification: "targeted fortification" based on analyses of breast milk proteins, and "adjustable fortification" based on the blood urea nitrogen (BUN) - reflected metabolic response of infants (10, 12). Despite these developments, there is still no consensus on the optimum fortification method; many different protocols are applied in NICUs worldwide (20, 21).

To the best of the investigators knowledge, no study has yet compared these two individualized fortification methods for nutrition of preterm infants. Therefore, the investigators compared the effects of targeted and adjustable protein fortification on the early growth of breastfed VLBW preterm infants.

ELIGIBILITY:
Inclusion Criteria:

- Very-low-birth-weight preterm infants ≤ 32 weeks of gestational age who were fed exclusively fortified breast milk.

Exclusion Criteria:

* The exclusion criteria were any congenital abnormality, a metabolic disease, necrotizing enterocolitis, bronchopulmonary dysplasia, and feeding with formula or formula plus breast milk.

Ages: 25 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very-low-birth-weight preterm infants ≤ 32 weeks of gestational age were included in the study and randomized into two groups according to the method of breast milk fortification.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Weight gain | 4 weeks
  The mean of weight gain (g/kg/day)
Head circumference | 4 weeks
  The mean of head circumference (mm/week)
Length | 4 weeks
  The mean of length (mm/week)

SECONDARY OUTCOMES:
Blood Urea Nitrogen (BUN) | 4 weeks
  The mean of BUN (mg/dL)
Albumin | 4 weeks
  The mean of albumin (g/dL)
Base deficit | 4 weeks
  The mean of base deficit (mEq/L)
Protein content | 4 weeks
  The mean of total daily intake of protein (g/kg/day)
Calorie intake | 4 weeks
  The mean of total daily intake of calorie (kcal/kg/day)
Carbonhydrate content | 4 weeks
  The mean of total daily intake of carbohydrate (g/kg/day)
Lipid content | 4 weeks
  The mean of total daily intake of lipid (g/kg/day)
Protein/Energy Ratio | 4 weeks
  The mean of total daily intake of Protein\Energy Ratio

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Ince, Prof., Study Director — Istanbul University

IPD SHARING:
Plan to Share IPD: Undecided
I'm not currently clear about sharing IPD. I will consider this at a later stage.